CLINICAL TRIAL: NCT05078177
Title: Trial of the Efficacy and Safety of Pathogenetic Therapy of Multiple Sclerosis and Other Autoimmune Diseases Using Intrathecal Rituximab
Brief Title: Safety and Efficacy of Intrathecal Rituximab in Patients With Multiple Sclerosis
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: St. Petersburg State Pavlov Medical University (Other)
Responsible Party: Principal Investigator, Ivan S Moiseev, Vice-director for science of R.M. Gorbacheva Memorial Institute of Hematology, Oncology and Transplantation, St. Petersburg State Pavlov Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: intrathecal_rtx_ms
Record Dates: First submitted 2021-10-01; First posted 2021-10-14 (Actual); Last update posted 2021-10-14 (Actual); Status verified 2021-10

CONDITIONS: Multiple Sclerosis
Keywords: Autoimmune Diseases; Rituximab
MeSH Terms: conditions — Multiple Sclerosis; Autoimmune Diseases | interventions — Rituximab; Reditux

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- AHSCT + intrathecal Rituximab (Experimental): AHSCT with reduced intensity condition regimen (RIC). Lumbar puncture with intrathecal injection of 25 mg Rituximab will be performed once from about D+12 to D+14 AHSCT, depending on the duration of cytopenia.
  Interventions: Drug: Rituximab

INTERVENTIONS:
Drug: Rituximab — All patients receive AHSCT with RIC (Cyclophosphamide, Antithymocyte globulin/Rituximab). After resolution of cytopenia (approximately from about D+12 to D+14 AHSCT), patients will receive intrathecal Rituximab.
  Other Names: Mabthera; Reditux; Acellbia

SUMMARY:
Considering the accumulated data on the pathogenesis of multiple sclerosis, indicating a significant role of B cells in the progression of the disease, the use of monoclonal antibodies to CD20 antigen, administered intrathecally to achieve adequate B-lymphodepletion in the barrier tissues can increase the duration of the recurrence-free course of autoimmune diseases, suspend their progression, and also prevent clinical relapse when memory B cells are detected.

DETAILED DESCRIPTION:
Multiple sclerosis (MS) is a chronic progressive autoimmune-mediated inflammatory demyelinating disease of the central nervous system (CNS), clinically manifested by impaired sensory motor function and cognitive impairment. In the pathogenesis of MS, T-cells make the main contribution to the process of inflammatory demyelination; however, the accumulated data on the pathogenesis of MS indicate a significant role of B cells in the progression of the disease. In addition to differentiation into plasma cells that produce autoantibodies, B lymphocytes stimulate T cell activity through antigen presentation, production of proinflammatory cytokines that trigger demyelination and differentiation into memory B cells that promote CD4 + T cell autoproliferation. The presence of "oligoclonal bands" in cerebrospinal fluid and demyelination plaques of brain tissue in MS patients is the result of persistent intrathecal clonal expansion of various B cell populations that contribute to the production of autoreactive antibodies. Thus, B cells located in the central nervous system, protected by the blood-brain barrier (BBB) and, as a consequence, not undergoing complete eradication due to limited penetration of the BBB by immunosuppressive drugs, are a potential target for the treatment of patients with MS. Depletion of B cells through the use of monoclonal antibodies to the CD20 antigen, which is expressed predominantly on mature B lymphocytes, is a promising direction in the therapy of autoimmune diseases. The most readily available anti-CD20 monoclonal antibody is rituximab. The available data from numerous studies on the use of intravenous rituximab have demonstrated a decrease in MR activity and clinical activity in patients with RRMS. At the same time, rituximab does not affect clinical outcomes in patients with PPMS and SPMS with a long history of the disease, probably due to insufficient antibody concentration in intact BBB in the CNS tissue affected by tertiary lymphoid follicles, because the ratio of rituximab concentration in CSF and serum after intravenous infusion ranges from 0.1% to 1-1.7%. Thus, to ensure a sufficient therapeutic concentration of rituximab in the tissues of the central nervous system, the use of the intrathecal route of drug administration is justified. To date, sufficient data have been accumulated on the safety of using intrathecal rituximab in the treatment of both oncological and autoimmune diseases (including MS).

Thus, the use of an anti-CD20 monoclonal antibody injected intrathecally in order to achieve adequate B-lymphodepletion in the barrier tissues can increase the duration of the recurrence-free course of autoimmune diseases, suspend their progression, and also prevent clinical relapse when memory B cells are detected.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65;
* 1.0-7.5 points on the EDSS scale (for MS);
* Length of illness - any;
* Disease progression during the last 6 months while taking drugs of 1st and 2nd lines;
* An established and confirmed diagnosis of an autoimmune disease in the previous stages of treatment;
* Ineffectiveness, inaccessibility or intolerance of Disease-Modifying Therapies;
* Relapse after AHSCT.
* Absence of severe concomitant somatic pathology;
* Left ventricular injection fraction > 50%;
* Karnofsky Performance Score (KPS) > 30%;
* The ability to take oral medications;
* Life expectancy is more than 1 month;
* Signed informed consent of the patient or legal representatives.

Exclusion Criteria:

* Moderate or severe cardiac dysfunction, left ventricular ejection fraction <50%
* Moderate or severe decrease in pulmonary function, FEV1 <70% or DLCO<70% of predicted
* Respiratory distress >grade I
* Severe organ dysfunction: AST or ALT >5 upper normal limits, bilirubin >1.5 upper normal limits, creatinine >2 upper normal limits
* Creatinine clearance < 60 mL/min
* Uncontrolled bacterial or fungal infection at the time of enrollment
* Requirement for vasopressor support at the time of enrollment
* Karnofsky performans status <30%
* Pregnancy
* Somatic or psychiatric disorder making the patient unable to sign informed consent

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2020-12-21 (Actual); Primary Completion 2022-12-21 (Estimated); Study Completion 2024-12-21 (Estimated)

PRIMARY OUTCOMES:
Multiple sclerosis progression free survival | 365 days
  To evaluate safety and effectiveness of intrathecal Rituximab in patients with refractory multiple sclerosis after AHSCT. Multiple sclerosis progression free survival

SECONDARY OUTCOMES:
Overall survival | 365 days
  To evaluate overall survival after AHSCT in combination with intrathecal Rituximab in patients with autoimmune diseases.
To evaluate adverse effects after intrathecal Rituximab | 365 days
  Toxicity based NCI CTCAE ver.5.0, including analysis of severe bacterial, fungal and viral infections incidence
Quality of life status 1 | 365 days
  Multiple sclerosis-specific questionnaire - HADS (Hospital Anxiety and Depression Scale) before and after AHSCT:
  0-7 points - normal; 8-10 - subclinically expressed anxiety/depression; 11-21 - clinically expressed anxiety/depression.
Quality of life status 2 | 365 days
  Multiple sclerosis-specific questionnaire - The Short Form-36 (SF-36) before and after AHSCT:
  The SF-36 consists of 36 questions grouped into eight scales: physical functioning, role-physical functioning, bodily pain, general health, vitality, social functioning, role-emotional, and mental health. The indicators of each scale are compiled in such a way that the higher the value of the indicator (from 0 to 100), the better the score on the chosen scale. Of these, two parameters are formed: the psychological and physical components of health.
Quality of life status 3 | 365 days
  Multiple sclerosis-specific questionnaire - Multiple Sclerosis Impact Scale (MSIS-29) before and after AHSCT:
  The MSIS-29 scale consists of 29 items and includes indicators observed over the previous two weeks, including 20 of which characterize physical condition, coordination and mobility, and 9 questions reflect the patient's mental state. Answers are ranked on a 5-point Likert scale from 1 to 5 (1 = none; 2 = little; 3 = moderate; 4 = significant; 5 = very strong) in one direction.
  The total score is the sum of all 29 responses and can range from 29 to 145. A higher score means a higher degree of disability. The result is assessed on a scale from 0 to 100, where a higher result means worse health.
Quality of life status 4 | 365 days
  Multiple sclerosis-specific questionnaire - Functional Assessment of Multiple Sclerosis (FAMS) before and after AHSCT:
  FAMS Total score (range=0-176) is derived by adding: 1) Mobility (r=0-28). 2) Symptoms (r=0-28). 3) Emotional well-being (r=0-28). 4) General contentment (r=0-28). 5) Thinking and fatigue (r=0-36). 6) Family/social wellbeing (r=0-28).
  Higher scores indicate better quality of life.
Neurological status 1 | 365 days
  Multiple sclerosis-specific questionnaire - EDSS (Expanded Disability Status Scale) before and after AHSCT:
  0 points - Normal neurologic exam; 1.0-1.5 - No disability, minimal signs in one or two Functional Systems (FS); 2.0-2.5 - Minimal disability in one or two FS; 3.0-3,5 - Moderate disability in one FS, fully ambulatory; 4.0-4.5 - Fully ambulatory without aid. Able to walk without aid or rest some 500 or 300 meters; 5.0-5.5 - Ambulatory without aid or rest for about 200 or 100 meters; 6.0 - Intermittent assistance required to walk about 100 meters; 6.5 - Constant bilateral assistance required to walk about 20 meters; 7.0-7.5 - Unable to walk beyond about 5 meters or more than a few steps; 8.0 - Essentially restricted to bed, but may be out of bed itself; 8.5 - Essentially restricted to bed; 9.0 - Helpless bed patient; can communicate and eat; 9.5 - Totally helpless bed patient; unable to communicate effectively or eat/swallow; 10 - Death due to MS
Evaluation of Immune system reconstitution after AHSCT 1 | 365 days
  Determination of absolute and relative values of the subpopulation composition of T-lymphocytes (CD3, CD4, CD8, CD45) and the ratio of T-helpers/T-cytotoxic cells before and after AHSCT.
Evaluation of Immune system reconstitution after AHSCT 2 | 365 days
  Determination of the absolute and relative number of CD19 + B-lymphocytes and analysis of subpopulations of B-lymphocytes: B1-cells (CD19+CD5+), B-2 cells (CD19+CD5-), memory B-cells (CD19+CD5-CD27+) before and after AHSCT.
Impact of autoHSCT+intrathecal Rituximab on brain structure anatomy | 365 days
  MRI 3,0 T

CONTACTS AND LOCATIONS:
Overall Officials: Ivan S Moiseev, MD, Ph.D, Principal Investigator — Pavlov First Saint Petersburg State Medical University
Locations (1):
- First Pavlov State Medical University of St. Petersburg, Saint Petersburg, Russia